CLINICAL TRIAL: NCT00088764
Title: Disclosure and Skills Training for Rheumatoid Arthritis
Brief Title: Pain and Stress Management for People With Rheumatoid Arthritis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Wayne State University (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Principal Investigator, Mark A. Lumley, Professor, Wayne State University
Allocation: Randomized | Model: Factorial | Masking: None
Other Study IDs: NIAMS-122; R01AR049059 (NIH); 1R01AR049059 (NIH)
Record Dates: First submitted 2004-08-04; First posted 2004-08-05 (Estimated); Last update posted 2013-08-15 (Estimated); Status verified 2013-08

CONDITIONS: Rheumatoid Arthritis
Keywords: Stress; Coping; Expressive Writing; Self-Efficacy; Disclosure
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Education: Either coping skills training or arthritis education interventions
  Interventions: Behavioral: Coping skills training; Behavioral: Arthritis education
- 2 (Experimental): Writing: Either emotional disclosure writing or health behavior writing
  Interventions: Behavioral: Written emotional disclosure; Behavioral: Health behavior writing

INTERVENTIONS:
Behavioral: Coping skills training — 8 sessions of pain and stress coping skills training
  Arms: 1
Behavioral: Written emotional disclosure — 4 sessions of writing about stress
  Arms: 2
Behavioral: Arthritis education — 8 sessions of learning about rheumatoid arthritis
  Arms: 1
Behavioral: Health behavior writing — 4 sessions of writing about various health behaviors
  Arms: 2

SUMMARY:
Self-management of rheumatoid arthritis (RA) symptoms using written emotional disclosure (ED), coping skills training (CST), or a combination of both may benefit people with RA. The purpose of this study is to determine the benefits of ED, CST, or CST and ED together in adults with RA. This study will be conducted at Wayne State University in Detroit, Michigan and Duke University Medical Center in Durham, North Carolina.

DETAILED DESCRIPTION:
Two self-management strategies hold promise for improving the health of people with RA: ED (writing about stress, RA, and coping options) and CST (learning six pain and stress coping skills). A strategy integrating ED with CST may be more effective than either intervention alone. This study will compare the effectiveness of ED, CST, ED in combination with CST, and control groups in alleviating the symptoms of RA.

This study will last until May 2009. Participants with RA will be randomly assigned to 1 of 4 treatment groups. Each participant will receive 3 writing sessions and 8 training sessions. Group 1 will receive ED writing followed by CST; Group 2 will receive ED writing followed by arthritis education; Group 3 will receive health behavior writing followed by CST; and Group 4 will receive health behavior writing followed by arthritis education.

Participants will be evaluated at baseline and at Months 1, 4, and 12 for pain, physical disability, psychological impairment, and disease activity. In addition, participants will record daily diaries for 30 days regarding their pain, symptoms, coping, stress, and mood prior to each of the evaluations. Changes in health status over time will be compared among groups.

ELIGIBILITY:
Inclusion Criteria:

* Meet American College of Rheumatology (ACR) 1987 criteria for RA

Exclusion Criteria:

* Other disorders that would significantly affect function (e.g., lupus, chronic obstructive pulmonary disease [COPD], congestive heart failure [CHF], cancer)
* Judged by the physician to have cognitive impairment (dementia, retardation, psychosis) or illiteracy
* Has experienced recent (last 6 months) significant stressor resulting in substantial emotional instability
* Currently in psychotherapy or a formal behavioral pain management program
* Unable to walk. Participants who use walking aids are not excluded.
* Physically unable to write

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Actual)
Dates: Start 2005-02; Primary Completion 2009-04 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Joint count | one year

SECONDARY OUTCOMES:
Psychological impairment | one year
Pain | one year
Physical disability | one year
C-reactive protein | one year
Fatigue | one year

CONTACTS AND LOCATIONS:
Overall Officials: Mark A. Lumley, PhD, Principal Investigator — Wayne State University
Locations (2):
- United States (2):
  - Wayne State University, Detroit, Michigan
  - Duke University Medical Center, Durham, North Carolina

REFERENCES:
- [Background] Kelley JE, Lumley MA, Leisen JC. Health effects of emotional disclosure in rheumatoid arthritis patients. Health Psychol. 1997 Jul;16(4):331-40. doi: 10.1037//0278-6133.16.4.331. PMID 9237085
- [Derived] Somers TJ, Shelby RA, Keefe FJ, Godiwala N, Lumley MA, Mosley-Williams A, Rice JR, Caldwell D. Disease severity and domain-specific arthritis self-efficacy: relationships to pain and functioning in patients with rheumatoid arthritis. Arthritis Care Res (Hoboken). 2010 Jun;62(6):848-56. doi: 10.1002/acr.20127. PMID 20535796